CLINICAL TRIAL: NCT00623714
Title: A Randomized, Placebo-Controlled, Crossover Study to Assess the Effects of Inhaled Fluticasone on Markers of Inflammation After Allergen Challenge in Patients With Allergic Asthma
Brief Title: Induced Sputum Study (0000-065)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-065; 065; 2008_509
Record Dates: First submitted 2008-02-11; First posted 2008-02-26 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental): study medication + Pbo
  Interventions: Drug: Comparator: fluticasone; Drug: Placebo
- Arm 2 (Experimental): Pbo + study medication
  Interventions: Drug: Comparator: fluticasone; Drug: Placebo

INTERVENTIONS:
Drug: Comparator: fluticasone — Two puffs, of 250 µg each, will be administered to each patient to obtain a 500-µg dose at each prespecified time point. A total of five (5) doses (500 µg) each of inhaled fluticasone will be administered in a 3-day period during Periods 1 and 2. Dosing will be twice a day for 3 days, ending after the morning dose on the third day.
  Other Names: fluticasone
Drug: Placebo — Two puffs, of placebo, will be administered to each patient at each prespecified time point. A total of five (5) doses of placebo will be administered during the single blind run-in phase. and matching placebo will be administered in a 3-day period during Periods 1 and 2. Dosing will be twice a day for 3 days, ending after the morning dose on the third day.

SUMMARY:
The primary goals of this study will be to implement innovative processing and detection assays to qualify induced sputum measurements of markers of allergen-induced airway inflammation. The results of this study are intended to form a platform to be used in the clinical development of novel asthma therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of mild to moderate persistent allergic asthma for at least 6 months with typical symptoms, including cough, wheezing, and shortness of breath, is clinically stable and has no history of recent respiratory tract infection within 3 weeks of the start of the study
* Patient, aside history of asthma, is judged to be in good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests.
* Patient is able to perform reproducible pulmonary function test.
* Patient has an allergic response to house dust mite allergen, demonstrates a positive early and late phase response to an inhaled allergen challenge (as defined by a bronchoconstrictive response)
* Patient is a nonsmoker for at least 12 months. Patients must have less than or equal to 10 pack years of smoking to be included. (10 pack years = one pack per day for 10 years.) Patients who have discontinued smoking for at least 10 months may be enrolled at the discretion of the investigator
* Patient is willing to avoid strenuous physical activity (i.e., strenuous or unaccustomed weight lifting, running, bicycling, etc.) for 72 hours prior to each visit when laboratory safety tests are obtained and 48 hours prior to allergen challenge

Exclusion Criteria:

* Patient has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses additional risk to the patient by their participation in the study
* Patient has taken oral corticosteroids within 8 weeks or inhaled corticosteroids/nasal corticosteroids within 4 weeks of screening and/or during the study
* Patient has a history of stroke, chronic seizures, or major neurological disorder
* Patient has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory (other than asthma), or genitourinary abnormalities or diseases, or has a history of neoplastic disease
* Patient is unable to refrain from or anticipates the use of any medication other than the ones permitted in this study, including prescription and non-prescription drugs or herbal remedies prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods), until the poststudy visit
* Patient consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages per day or >21 drink equivalents per week.
* Patient consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, or other caffeinated beverages per day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered: 28-Jan-2008
  Last Patient, Last Visit: 05-Mar-2009
  1 site
Pre-assignment Details: Inclusion
  * Mild/moderate allergic asthma
  * Allergic to house, dust, mite allergen
  * Early and late allergic response to inhaled allergen challenge
  Randomized sequence of treatments including 500 μg fluticasone or placebo in treatment periods 1 & 2. Treatment was twice a day (b.i.d.) for total of 5 doses over 3-day period.
Groups:
- Placebo Then Fluticasone: Days 1-2 Placebo twice a Day (b.i.d.) + Day 3 Placebo single dose, Days 1-2 500 µg Fluticasone b.i.d. + Day 3 500 µg Fluticasone single dose
- Fluticasone Then Placebo: Days 1-2 500 µg Fluticasone b.i.d. + Day 3 500 µg Fluticasone single dose, Days 1-2 Placebo b.i.d. + Day 3 Placebo single dose
Period: Period 1
Arm/Group | Placebo Then Fluticasone | Fluticasone Then Placebo
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Placebo Then Fluticasone | Fluticasone Then Placebo
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All Randomized Patients
Arm/Group | All Patients
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 25.9 [21 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Hour 24 Fold Change From Period Baseline in Interleukin-5 (IL-5) Protein Concentration (pg/mL)
Time Frame: Baseline and 24 hours post allergen challenge
Population: All Patients as Treated
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Placebo: Days 1-2 Placebo b.i.d. + Day 3 Placebo single dose
- Fluticasone: Days 1-2 500 µg Fluticasone b.i.d. + Day 3 500 µg Fluticasone single dose
Arm/Group | Placebo | Fluticasone
Number analyzed (Participants) | 13 | 13
pg/mL | 2.57 [1.37 to 4.84] | 0.87 [0.46 to 1.64]
Statistical Analysis 1: Comparison: Placebo vs Fluticasone; Test type: Superiority or Other; p = 0.011, ANOVA — 1-sided, alpha = 0.05; Analysis performed on log-transformed fold change from baseline and results were back-transformed for reporting; Geometric Mean Fold Difference = 0.34, 90% CI 2-sided [0.16 to 0.70]

2. Secondary Outcome: Hour 24 Fold Change From Period Baseline in Interleukin-13 (IL-13) Protein Concentration (pg/mL)
Time Frame: Baseline and 24 hours post allergen challenge
Population: All Patients as Treated
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Placebo | Fluticasone
Number analyzed (Participants) | 13 | 13
pg/mL | 2.11 [1.41 to 3.17] | 0.85 [0.57 to 1.28]
Statistical Analysis 1: Comparison: Placebo vs Fluticasone; Test type: Superiority or Other; p = 0.002, ANOVA — 1-sided, alpha = 0.05; Analysis performed on log-transformed fold change from baseline and results were back-transformed for reporting; Geometric Mean Fold Difference = 0.40, 95% CI 2-sided [0.26 to 0.63]

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected from the time the consent is signed through the 14 day follow up period after all treatment periods were completed
Description: AE s were assessed by clinical evaluation including vital signs, physical examination, medical history, clinical laboratory safety assessment (hematology, chemistry, urinalysis), and ECG at timepoints specified in the study. Patients were queried at each visit for any adverse experiences since the previous visit.
Arm/Group | Placebo | Fluticasone
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 5/13 | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Fluticasone (N=13)
Fatigue (General disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Muscle Contractions Involuntary (Nervous system disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.